CLINICAL TRIAL: NCT05298605
Title: Faith in Action! A Cluster-Randomized Trial to Evaluate the Efficacy of a Church-based Navigation Model to Increase Breast Cancer Screening Among Korean Women in Los Angeles
Brief Title: Faith in Action! A Church-Based Navigation Model to Increase Breast Cancer Screening in Korean Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: California Breast Cancer Research Program (Other)
Responsible Party: Principal Investigator, Robert Haile, Director, Cancer Research Center for Health Equity, Professor, Department of Medicine, Associate Director for Population Health, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00001641
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Female; Health Knowledge, Attitudes, Practice; Cancer Screening; Health Disparities
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faith in Action! (Experimental): A train-the-trainer approach will be used to educate lay health navigators to present the culturally adapted "Faith in Action!" curriculum and to provide breast cancer screening navigation to Korean American women within faith-based settings
  Interventions: Behavioral: Faith in Action! Church-based Navigation Model
- Control (Active Comparator): A presentation of lifestyle recommendations (e.g., physical activity, nutrition) will be provided to control groups.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Faith in Action! Church-based Navigation Model — Cancer screening education and navigation by identified trained navigators in faith based settings + American Cancer Society Screening Guidelines pamphlet
  Arms: Faith in Action!
Other: Control — Presentation on healthy behaviors (physical activity, nutrition) + American Cancer Society Screening Guidelines pamphlet
  Arms: Control

SUMMARY:
The purpose of this research is to develop a culturally adapted "Faith in Action!" curriculum to train lay health navigators to provide breast cancer screening navigation to Korean American women within faith-based settings and evaluate whether the culturally adapted "Faith in Action!" curriculum increases adherence to breast cancer screening guidelines among Korean American women within faith-based settings in Los Angeles, California. The primary research procedures include trainings and key informant interviews with lay health navigators in faith-based settings followed by a cluster randomized trial to evaluate the intervention.

DETAILED DESCRIPTION:
A parallel cluster randomized trial (CRT) with staggered roll-out will be conducted to evaluate the efficacy of the "Faith in Action!" intervention on breast cancer screening rates among Korean American women. This will involve two blocks of 8 churches each (total 16 churches) randomized to either the intervention or waitlist control.

A train the trainer approach will be used to educate and certify lay health navigators identified by targeted Korean church leaders from selected churches. The trained health navigators will be deployed back to the churches and community settings with tools and resources to deliver cancer education and increase motivation to participate in breast cancer screening through proven approaches such as one-on-one education, small media and workshops.

The research objectives are to:

1. Develop a culturally adapted "Faith in Action!" curriculum to train lay health navigators to provide breast cancer screening navigation to Korean American women within faith-based settings.
2. Evaluate whether the culturally adapted "Faith in Action!" curriculum increases adherence to breast cancer screening guidelines among Korean American women within faith-based settings.

It is hypothesized that the implementation of this culturally adapted cancer screening training curriculum for lay health navigators, built upon the Korean communities' frequent engagement with "expert" schools and deployed among existing networks in the faith-based Korean community, will increase adherence to breast cancer screening guidelines among underserved Korean American women.

ELIGIBILITY:
Inclusion Criteria:

* Korean woman who is 45 years or older
* Does not currently have a breast cancer diagnosis
* Non-adherent to cancer screening (did not receive mammogram in last 2 years based on self-report)
* Prospective or current member of participating Korean Churches
* Willing to participate in study

Exclusion Criteria:

* Does not meet inclusion criteria as described above

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women at risk of breast cancer
Enrollment: 320 (Estimated)
Dates: Start 2022-07-16 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Screening adherence | up to 6 months from end of program
  Percent change in adherence to breast cancer screening guidelines within 6 months from end of program

SECONDARY OUTCOMES:
Breast Cancer Screening Beliefs (Knowledge, Perception, and perceived risk) | up to 6 months
  Assessed in validated, Breast Cancer Screening Beliefs Questionnaire (Kwok et al) including Likert-type questions (13 items and 3 sub scales, items range 1-5, strongly agree to strongly disagree)
Participant knowledge, attitudes, and beliefs towards screening (Qualitative) | up to 6 months
  Assessed in qualitative interviews
Change in Knowledge of Breast Cancer Screening | up to 6 months
  Knowledge of breast cancer screening based on pre-post knowledge assessments adapted Cancer 101 assessments (3 knowledge assessments (5 items each), response categories: Agree, Disagree, or Unsure).

OTHER OUTCOMES:
Change in NIH PROMIS Global Health | Up to 6 months
  Change in continuous NIH PROMIS converted T-Scores (mean 50, SD:10) at 6 months. Questionnaire includes physical and mental health domains (4 items total, likert 5-point scale, converted to continuous T scores)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Kaiser Permanente Center for Health Equity, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
Aggregated data at cluster level will be available upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Within one year from end of study
Access Criteria: Published protocol and uploaded to ClinicalTrials.Gov.

REFERENCES:
- [Derived] Gresham G, Kim DH, Sung MJ, Diniz MA, Finster L, Fine M, Jeon C, Herrmann AK, Lee JY, Surani Z, Haile RW. Protocol for a cluster randomized trial to evaluate a faith-based breast cancer screening navigation model. Trials. 2026 Jan 29. doi: 10.1186/s13063-025-09397-2. Online ahead of print. PMID 41612469